CLINICAL TRIAL: NCT03794544
Title: A Phase 2 Open-label, Multicenter, Randomized, Multidrug Platform Study of Neoadjuvant Durvalumab Alone or in Combination With Novel Agents in Subjects With Resectable, Early-stage (I [> 2 cm] to IIIA) Non-small Cell Lung Cancer (NeoCOAST)
Brief Title: Neoadjuvant Durvalumab Alone or in Combination With Novel Agents in Resectable Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9108C00002
Record Dates: First submitted 2018-12-10; First posted 2019-01-07 (Actual); Results first posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Resectable; Early-stage; NSCLC
Keywords: Neoadjuvant; Non-small Cell Lung Cancer; Cancer; Lung; Resectable; Early-stage; Stage I; Stage II; Stage IIIA; Durvalumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — durvalumab; monalizumab; danvatirsen

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled and randomized into a durvalumab monotherapy arm or into a durvalumab plus other novel therapy arms. Up to approximately 25 sites globally will participate in this study. New treatment arms may be added in the future. Participants will be treated with a single durvalumab dose alone or in combination with other agents. After the single cycle treatment period participants will have the standard surgical resection planned. All participants will have a post-resection monitoring visit. Study treatment will be discontinued upon disease progression, unacceptable toxicity, or other investigators' reasons.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Durvalumab 1500 mg (Experimental): Participants will receive durvalumab 1500 mg intravenously (IV) every 4 weeks (Q4W; on Week 1 Day 1) until disease progression, unacceptable toxicity, or other reason of treatment discontinuation over a 28-day treatment period. Surgical resection will be planned between Day 29 and Day 42. After surgical resection, participants will be followed up to Day 105 (starting from Week 1 Day 1).
  Interventions: Drug: Durvalumab
- Durvalumab 1500 mg + Oleclumab 3000 mg (Experimental): Participants will receive durvalumab 1500 mg IV Q4W (on Week 1 Day 1) and oleclumab 3000 mg IV every 2 weeks (Q2W; on Week 1 Day 1 and Week 3 Day 1) until disease progression, unacceptable toxicity, or other reason of treatment discontinuation over a 28-day treatment period. Surgical resection will be planned between Day 29 and Day 42. After surgical resection, participants will be followed up to Day 105 (starting from Week 1 Day 1).
  Interventions: Drug: Durvalumab; Combination Product: Oleclumab
- Durvalumab 1500 mg + Monalizumab 750 mg (Experimental): Participants will receive durvalumab 1500 mg IV Q4W (on Week 1 Day 1) and monalizumab 750 mg IV Q2W (on Week 1 Day 1 and Week 3 Day 1) until disease progression, unacceptable toxicity, or other reason of treatment discontinuation over a 28-day treatment period. Surgical resection will be planned between Day 29 and Day 42. After surgical resection, participants will be followed up to Day 105 (starting from Week 1 Day 1).
  Interventions: Drug: Durvalumab; Combination Product: Monalizumab
- Durvalumab 1500 mg + Danvatirsen 200 mg (Experimental): Participants will receive danvatirsen 200 mg IV on Days 1, 3, and 5 of Week 0 (7-day danvatirsen lead-in period), followed by durvalumab 1500 mg IV Q4W (on Week 1 Day 1) and danvatirsen 200 mg IV every week (on Week 1 Day 1, Week 2 Day 1, Week 3 Day 1, and Week 4 Day 1) until disease progression, unacceptable toxicity, or other reason of treatment discontinuation over a 28-day treatment period. Surgical resection will be planned between Day 29 and Day 42. After surgical resection, participants will be followed up to Day 105 (starting from Week 1 Day 1).
  Interventions: Drug: Durvalumab; Combination Product: Danvatirsen

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500 mg IV will be administered Q4W (on Week 1 Day 1) until disease progression, unacceptable toxicity, or other reason of treatment discontinuation over a 28-day treatment period.
  Other Names: MEDI4736
Combination Product: Oleclumab — Oleclumab 3000 mg IV will be administered Q2W (on Week 1 Day 1 and Week 3 Day 1) until disease progression, unacceptable toxicity, or other reason of treatment discontinuation over a 28-day treatment period.
  Other Names: MEDI9447
  Arms: Durvalumab 1500 mg + Oleclumab 3000 mg
Combination Product: Monalizumab — Monalizumab 750 mg IV will be administered Q2W (on Week 1 Day 1 and Week 3 Day 1) until disease progression, unacceptable toxicity, or other reason of treatment discontinuation over a 28-day treatment period.
  Other Names: IPH2201
  Arms: Durvalumab 1500 mg + Monalizumab 750 mg
Combination Product: Danvatirsen — Danvatirsen 200 mg IV will be administered on Days 1, 3, and 5 of Week 0 (7-day danvatirsen lead-in period) and later every week (on Week 1 Day 1, Week 2 Day 1, Week 3 Day 1, and Week 4 Day 1) until disease progression, unacceptable toxicity, or other reason of treatment discontinuation over a 28-day treatment period.
  Other Names: AZD9150
  Arms: Durvalumab 1500 mg + Danvatirsen 200 mg

SUMMARY:
Study D9108C00002 (NeoCOAST) is a platform study assessing the effectiveness and safety of neoadjuvant durvalumab alone or in combination with novel agents in participants with resectable, early-stage (Stage I [>2cm] to IIIA) non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically and/or histologically-documented NSCLC

   1. Stage I (> 2 cm) to IIIA (for participants with N2 disease, only those with 1 single nodal station ≤ 3 cm are eligible) NSCLC according to the 8th edition of American Joint Committee on Cancer staging classification
   2. Amenable to complete surgical resection
   3. Have not received any other therapy for this condition
2. Predicted forced expiratory volume in one second (FEV1) ≥ 50%
3. Predicted diffusing capacity of the lungs for carbon monoxide (DLCO) ≥ 50%
4. ECOG 0 or 1
5. Adequate organ function

Exclusion Criteria:

1. Participants with small-cell lung cancer or mixed small-cell lung cancer
2. Participants who require or may require pneumonectomy
3. Prior treatment with programmed cell death ligand-1 (PD-L1), PD-L1, or cytotoxic T-lymphocyte antigen 4 (CTLA-4) inhibitors
4. Current or prior use of immunosuppressive medication within 14 days before the first dose of study drug.
5. Active or prior documented autoimmune or inflammatory disorders. The following are exceptions to this criterion:

   1. Participants with vitiligo or alopecia
   2. Participants with hypothyroidism on hormone replacement
   3. Any chronic skin condition that does not require systemic therapy
   4. Participants without active disease in the last 5 years may be included but only after consultation with the study physician
   5. Participants with celiac disease controlled by diet alone
6. Pregnant or breast-feeding female
7. Major surgical procedure within prior 30 days
8. History of active primary immunodeficiency
9. Active infection including tuberculosis, hepatitis B, hepatitis C, or HIV
10. QTc interval (QTc) ≥ 470 ms
11. Uncontrolled intercurrent illness that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the participant to give written informed consent
12. Receipt of live attenuated vaccination within 30 days prior to study entry
13. History of another primary malignancy except for:

    1. Curative-treated malignancy with no known active disease > 2 years before enrollment on the study
    2. Curative-treated non-melanoma skin cancer and/or carcinoma in-situ

Ages: 18 Years to 102 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (10):
  - Research Site, La Jolla, California
  - Research Site, Fort Myers, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Baltimore, Maryland
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
- Research Site, Montreal, Quebec, Canada
- France (2):
  - Research Site, Marseille
  - Research Site, Toulouse
- Research Site, Orbassano, Italy
- Research Site, Porto, Portugal
- Spain (2):
  - Research Site, A Coruña
  - Research Site, Barcelona
- Research Site, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Cascone T, Kar G, Spicer JD, Garcia-Campelo R, Weder W, Daniel DB, Spigel DR, Hussein M, Mazieres J, Oliveira J, Yau EH, Spira AI, Anagnostou V, Mager R, Hamid O, Cheng LY, Zheng Y, Blando J, Tan TH, Surace M, Rodriguez-Canales J, Gopalakrishnan V, Sellman BR, Grenga I, Soo-Hoo Y, Kumar R, McGrath L, Forde PM. Neoadjuvant Durvalumab Alone or Combined with Novel Immuno-Oncology Agents in Resectable Lung Cancer: The Phase II NeoCOAST Platform Trial. Cancer Discov. 2023 Nov 1;13(11):2394-2411. doi: 10.1158/2159-8290.CD-23-0436. PMID 37707791
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9108C00002&attachmentIdentifier=e88d14fa-1bd3-4d48-b0e5-6834aadf8fef&fileName=NeoCOAST_Protocol_Amd_2_redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9108C00002&attachmentIdentifier=4040b9c0-98e9-4de7-ac0d-a934f8c86908&fileName=d9108c00002-sap-ed4_redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9108C00002&attachmentIdentifier=0eea76d6-523a-4327-a88e-863b0e6531e4&fileName=Synopsis-NeoCOAST_Final_version_01Dec21-Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was interrupted due to COVID-19 pandemic from 13Apr2020 to 07May2020.
Groups:
- Durvalumab 1500 mg: Participants received durvalumab 1500 mg intravenously (IV) every 4 weeks (Q4W; on Week 1 Day 1) until disease progression, unacceptable toxicity, or other reason of treatment discontinuation over a 28-day treatment period. Surgical resection was planned between Day 29 and Day 42. After surgical resection, participants were followed up to Day 105 (starting from Week 1 Day 1).
- Durvalumab 1500 mg + Oleclumab 3000 mg: Participants received durvalumab 1500 mg IV Q4W (on Week 1 Day 1) and oleclumab 3000 mg IV every 2 weeks (Q2W; on Week 1 Day 1 and Week 3 Day 1) until disease progression, unacceptable toxicity, or other reason of treatment discontinuation over a 28-day treatment period. Surgical resection was planned between Day 29 and Day 42. After surgical resection, participants were followed up to Day 105 (starting from Week 1 Day 1).
- Durvalumab 1500 mg + Monalizumab 750 mg: Participants received durvalumab 1500 mg IV Q4W (on Week 1 Day 1) and monalizumab 750 mg IV Q2W (on Week 1 Day 1 and Week 3 Day 1) until disease progression, unacceptable toxicity, or other reason of treatment discontinuation over a 28-day treatment period. Surgical resection was planned between Day 29 and Day 42. After surgical resection, participants were followed up to Day 105 (starting from Week 1 Day 1).
- Durvalumab 1500 mg + Danvatirsen 200 mg: Participants received danvatirsen 200 mg IV on Days 1, 3, and 5 of Week 0 (7-day danvatirsen lead-in period), followed by durvalumab 1500 mg IV Q4W (on Week 1 Day 1) and danvatirsen 200 mg IV every week (on Week 1 Day 1, Week 2 Day 1, Week 3 Day 1, and Week 4 Day 1) until disease progression, unacceptable toxicity, or other reason of treatment discontinuation over a 28-day treatment period. Surgical resection was planned between Day 29 and Day 42. After surgical resection, participants were followed up to Day 105 (starting from Week 1 Day 1).
Period: Overall Study
Arm/Group | Durvalumab 1500 mg | Durvalumab 1500 mg + Oleclumab 3000 mg | Durvalumab 1500 mg + Monalizumab 750 mg | Durvalumab 1500 mg + Danvatirsen 200 mg
Started | 27 | 21 | 20 | 16
Treated | 26 | 21 | 20 | 16
Completed | 26 | 18 | 19 | 15
Not Completed | 1 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Other | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included participants who were randomized and were analyzed according to their randomized treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Durvalumab 1500 mg | Durvalumab 1500 mg + Oleclumab 3000 mg | Durvalumab 1500 mg + Monalizumab 750 mg | Durvalumab 1500 mg + Danvatirsen 200 mg | Total
Number analyzed (Participants) | 27 | 21 | 20 | 16 | 84
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.1 (9.0) | 65.5 (7.5) | 65.1 (6.3) | 72.9 (7.9) | 67.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 6 | 6 | 34
  Male | 14 | 12 | 14 | 10 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 2 | 3
  Not Hispanic or Latino | 26 | 21 | 20 | 14 | 81
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 0 | 5
  White | 23 | 20 | 19 | 13 | 75
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Major Pathological Response Rate
Description: Major pathological response rate is defined as percentage of participants with <=10% residual viable tumor cells in the resected specimen.
Time Frame: Day 1 through Day 42
Population: The ITT population included participants who were randomized and were analyzed according to their randomized treatment group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab 1500 mg | Durvalumab 1500 mg + Oleclumab 3000 mg | Durvalumab 1500 mg + Monalizumab 750 mg | Durvalumab 1500 mg + Danvatirsen 200 mg
Number analyzed (Participants) | 27 | 21 | 20 | 16
Percentage of participants | 11.1 [2.4 to 29.2] | 19.0 [5.4 to 41.9] | 30.0 [11.9 to 54.3] | 31.3 [11.0 to 58.7]

2. Secondary Outcome: Pathological Complete Response (pCR) Rate
Description: The pCR rate is defined as percentage of participants with no residual viable tumor cells in the resected specimen.
Time Frame: Day 1 through Day 42
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab 1500 mg | Durvalumab 1500 mg + Oleclumab 3000 mg | Durvalumab 1500 mg + Monalizumab 750 mg | Durvalumab 1500 mg + Danvatirsen 200 mg
Number analyzed (Participants) | 27 | 21 | 20 | 16
Percentage of participants | 3.7 [0.1 to 19.0] | 9.5 [1.2 to 30.4] | 10.0 [1.2 to 31.7] | 12.5 [1.6 to 38.3]

3. Secondary Outcome: Feasibility to Surgery
Description: Feasibility to surgery is defined as the percentage of participants who underwent the planned surgery within Days 29 to 42 after Week 1 Day 1.
Time Frame: Day 29 to Day 42 after Week 1 Day 1
Population: As-treated population included all participants who received any study drug and analyzed according to the treatment they actually received.
Measure: Number; unit: Percentage of participants
Arm/Group | Durvalumab 1500 mg | Durvalumab 1500 mg + Oleclumab 3000 mg | Durvalumab 1500 mg + Monalizumab 750 mg | Durvalumab 1500 mg + Danvatirsen 200 mg
Number analyzed (Participants) | 26 | 21 | 20 | 16
Percentage of participants | 84.6 [0.1 to 19.0] | 81.0 [1.2 to 30.4] | 90.0 [1.2 to 31.7] | 93.8 [1.6 to 38.3]

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: From Day 1 through Day 105
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab 1500 mg | Durvalumab 1500 mg + Oleclumab 3000 mg | Durvalumab 1500 mg + Monalizumab 750 mg | Durvalumab 1500 mg + Danvatirsen 200 mg
Number analyzed (Participants) | 26 | 21 | 20 | 16
Participants
  Any TEAEs | 18 | 19 | 15 | 13
  Any TESAEs | 3 | 2 | 1 | 5

5. Secondary Outcome: Number of Participants With Grade 3 or Grade 4 Clinical Laboratory Toxicities
Description: Participants with Grade 3 or Grade 4 clinical laboratory toxicities are reported. Laboratory tests included hematology, coagulation, chemistry, and urinalysis.
Time Frame: From Day 1 through Day 105
Population: As-treated population included all participants who received any study drug and analyzed according to the treatment they actually received. 'Number Analyzed' denotes the participants analyzed for the specified laboratory parameters.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab 1500 mg | Durvalumab 1500 mg + Oleclumab 3000 mg | Durvalumab 1500 mg + Monalizumab 750 mg | Durvalumab 1500 mg + Danvatirsen 200 mg
Number analyzed (Participants) | 26 | 21 | 20 | 16
Participants
  Alanine aminotransferase increased: number analyzed (Participants) | 25 | 21 | 20 | 16
  Alanine aminotransferase increased | 0 | 0 | 0 | 2
  Gamma glutamyl transferase increased: number analyzed (Participants) | 25 | 21 | 18 | 16
  Gamma glutamyl transferase increased | 0 | 0 | 0 | 1
  Lipase increased: number analyzed (Participants) | 25 | 21 | 19 | 16
  Lipase increased | 1 | 1 | 1 | 0
  Hyponatremia: number analyzed (Participants) | 25 | 21 | 20 | 16
  Hyponatremia | 2 | 0 | 0 | 0
  Lymphocyte count decreased | 0 | 0 | 0 | 1

6. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: Participants with abnormal vital sign reported as TEAEs are reported.
Time Frame: From Day 1 through Day 105
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab 1500 mg | Durvalumab 1500 mg + Oleclumab 3000 mg | Durvalumab 1500 mg + Monalizumab 750 mg | Durvalumab 1500 mg + Danvatirsen 200 mg
Number analyzed (Participants) | 26 | 21 | 20 | 16
Participants
  Palpitations | 1 | 0 | 0 | 0
  Pyrexia | 1 | 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 through Day 105
Description: As-treated population was considered for collecting AEs data. As-treated population included all participants who received any study drug and analyzed according to the treatment they actually received.
Arm/Group | Durvalumab 1500 mg | Durvalumab 1500 mg + Oleclumab 3000 mg | Durvalumab 1500 mg + Monalizumab 750 mg | Durvalumab 1500 mg + Danvatirsen 200 mg
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/21 | 0/20 | 1/16
Serious Adverse Events (participants affected / at risk) | 3/26 | 2/21 | 1/20 | 5/16
Other Adverse Events (participants affected / at risk) | 18/26 | 19/21 | 14/20 | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab 1500 mg (N=26) | Durvalumab 1500 mg + Oleclumab 3000 mg (N=21) | Durvalumab 1500 mg + Monalizumab 750 mg (N=20) | Durvalumab 1500 mg + Danvatirsen 200 mg (N=16)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal infarct (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab 1500 mg (N=26) | Durvalumab 1500 mg + Oleclumab 3000 mg (N=21) | Durvalumab 1500 mg + Monalizumab 750 mg (N=20) | Durvalumab 1500 mg + Danvatirsen 200 mg (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 6 (6) | 4 (4) | 2 (2) | 3 (3)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prothrombin time shortened (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tri-iodothyronine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest wall mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The pharmacokinetic and immunogenicity samples are still being analyzed. Results for these outcome measures will be posted by 30Jun2022.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT03794544/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT03794544/SAP_001.pdf